CLINICAL TRIAL: NCT01965119
Title: Pilot Study of Ruxolitinib in Relapsed or Refractory Hodgkin Lymphoma and Primary Mediastinal Large B-cell Lymphoma
Acronym: JAK2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, M.D., PhD., Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2013-06-039
Record Dates: First submitted 2013-10-09; First posted 2013-10-18 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma; Primary Mediastinal Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib (Experimental): 20 mg orally twice a day for 4 weeks (One cycle) Treatment continued until documented disease progression or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 20 mg orally twice a day for 4 weeks (One cycle) Treatment continued until documented disease progression or unacceptable toxicity.
  Other Names: jakavi

SUMMARY:
The purpose of this study is that ruxolitinib may be a possible treatment option for relapsed or refractory patients with Hodgkin and primary mediastinal large B-cell lymphoma.

DETAILED DESCRIPTION:
Patients will take ruxolitinib 20 mg orally twice a day, 40mg in total per day, for 4 weeks.4 weeks is 1 cycle. Treatment will be continued until documented disease progression or unacceptable toxicity and the maximum period of treatment is 16 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Hodgkin lymphoma or primary mediastinal large B-cell lymphoma
* Patient should belong to any one of following clinical situations A.Patient who are not able to get autologous stem cell transplantation after relapsing the salvage chemotherapy B. Relapsed after autologous stem cell transplantation C. Refractory to salvage chemotherapy or autologous stem cell transplantation
* Adequate organ function as defined by the following criteria:

A. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy B. Total serum bilirubin ≤1.5 x ULN C. Absolute neutrophil count (ANC) ≥ 1500/µL D. Platelets ≥ 100,000/µL E. Hemoglobin ≥ 9.0 g/dL (may be transfused or erythropoietin treated) F. Serum calcium ≤ 12.0 mg/dL G. Serum creatinine ≤ 1.5 x ULN

* At least one measurable lesion
* ECOG PS 0-2
* Informed consent
* Age from 19 to 80

Exclusion Criteria:

* Previously received allogeneic stem cell transplantation
* History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease or secondary CNS involvement on CT or MRI scan.
* Currently uncontrolled active infection
* Previous history of recurrent herpes zoster or recurrent tuberculosis
* Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
* Pregnant or lactating females or patients who ar not willing to use an adequate method of birth control for the duration of the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of disease control including complete response (CR), partial response (PR) and stable disease (SD) | From date of enrollment until the date first documented disease progression or unacceptable toxicity, whichever came first, assessed up to 48months

SECONDARY OUTCOMES:
Toxicity profile | from the date of informed consent signature to 30days after last drug administration
  CTCAE v4 (Common Terminology Criteria for Adverse Events v4.0) In the present study, toxicities will be recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Event (CTCAE), version 4.0. The full CTCAE documentation is available on the NCI web site, at the following address: http://ctep.cancer.gov/forms/CTCAEv4.pdf The occurrence of severe adverse event (SAE) should be also reported to the Novartis Safety Office within 24 hours.
Overal Survival | from the date of first drug administration until the date of death, assessed up to 48months

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, PhD, Principal Investigator — Samsung Medical Center
Locations (7):
- South Korea (7):
  - Busan University Hospital, Busan
  - Dong-A University, Busan
  - Kosin University Gospel Hospital, Busan
  - Asan Medical Center, Seoul
  - Korean Cancer Center Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Kim SJ, Yoon DH, Kang HJ, Hong JY, Lee HS, Oh SY, Shin HJ, Kong JH, Yi JH, Sakamoto K, Ko YH, Huh J, Lee SS, Takeuchi K, Shin DY, Suh C, Kim WS. Ruxolitinib shows activity against Hodgkin lymphoma but not primary mediastinal large B-cell lymphoma. BMC Cancer. 2019 Nov 10;19(1):1080. doi: 10.1186/s12885-019-6303-z. PMID 31707975